CLINICAL TRIAL: NCT04667429
Title: A Phase I,Double-Blind, Placebo-Controlled, Multiple Oral Dose, Safety, Tolerability, Pharmacokinetics and Food Effect Study of HEC83518 Tablets in Healthy Chinese Subjects
Brief Title: the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC83518 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC83518-P-02 / CRC-C2048
Record Dates: First submitted 2020-11-24; First posted 2020-12-14 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ascending Multiple Dose Study is Double-blind design; Food Effect Study is open-label design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Food effect (Experimental): HEC83518 40mg will be administered fasted, or with high-fat meal for once.
  Interventions: Other: Food
- Multiple Ascending Doses-HEC83518 20mg (Experimental): HEC83518 20mg will be administered before sleep for 15 days .
  Interventions: Drug: HEC83518
- Multiple Ascending Doses-HEC83518 40mg (Experimental): HEC83518 40mg will be administered before sleep for 15 days .
  Interventions: Drug: HEC83518
- Multiple Ascending Doses-HEC83518 80mg (Experimental): HEC83518 80mg will be administered before sleep for 15 days .
  Interventions: Drug: HEC83518
- Multiple Ascending Doses-placebo (Placebo Comparator): Placebo will be administered before sleep for 15 days .
  Interventions: Drug: placebo

INTERVENTIONS:
Other: Food — HEC83518 40mg will be taken orally fasted or with food
  Arms: Food effect
Drug: HEC83518 — HEC83518 will be taken orally before sleep for 15 days
  Arms: Multiple Ascending Doses-HEC83518 20mg; Multiple Ascending Doses-HEC83518 40mg; Multiple Ascending Doses-HEC83518 80mg
Drug: placebo — The placebo will be administered before sleep for 15 days.
  Arms: Multiple Ascending Doses-placebo

SUMMARY:
Multiple Dose Safety, Tolerability, PK ，PD and Food Effect Study of HEC83518 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
2. Without Plan for pregnancy or pregnant within 3 months after enrollment throughout the trial.
3. Subjects aged between 18 and 45 (both inclusive) years old.
4. Healthy volunteers have a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18 and ≤28 kg/m2 at screening.
5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. Subjects with a heart rate ≥100 beats per minute or ≤ 60 beats per minute at screening or baseline.
2. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
3. Subjects with history of digestive system,urinary system, liver,central nervous system, blood system, endocrine system,respiratory system,immune system,cardiovascular system,and/or malignant tumor or others medical conditions (such as history of mental illness, etc.) that are not suitable for clinical trial participation;Subjects with history of stroke, epilepsy, bipolar disorder/mania, high intraocular pressure, or acute angular-closure glaucoma.
4. Subjects with history of sleep-related illness.
5. Subjects with history of severe involuntary hypoglycemia
6. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s) ,or anaphylaxis physique.
7. Use of any prescription or non-prescription medications within 14 days prior to initial dosing,or Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.
8. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
9. Positive results from urine drug screen test.
10. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
11. Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug.
12. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
13. Subjects who plan to receive or have had organ transplants.
14. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential. 15 Subjects who participated in another clinical trial within 3 months prior to initial dosing.

16.Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Adverse event | up to 34 days
  To assess the safety and tolerability of therapy

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) from time zero to infinity(AUC0-∞ ) | up to 72 hours
Maximum Plasma Concentration ( Cmax) | up to 72 hours
Time to peak(tmax) | up to 72 hours
Apparent terminal elimination half-life(t½) | up to 72 hours
Apparent volume of distribution(Vz/F) | up to 72 hours
The Mean Residence Time#(MRT) | up to 72 hours
The Apparent Clearance (CL/F) | up to 72 hours
The Accumulation Ratio(R) | up to 60 hours
Food Effect on the Cmax | up to 72 hours
Food Effect on the AUC | up to 72 hours

OTHER OUTCOMES:
Karolinska sleepiness Scale（KSS） | up to 24 hour
  This is a 9-point scale (1 = extremely alert, 3 = alert, 5 = neither alert nor sleepy,7 = sleepy - but no difficulty remaining awake,and 9 = extremely sleepy - fighting sleep).The score of KSS scale will be recorded at different time and the change score compared with baseline will be analysed to evaluated the start of effective time, the most effective time and the recovered time to baseline.
Latency to sleep measured by a polysomnograph | during the sleep time on the night(from 22:00-22:30 to the next morning wake-up)
Wake After Sleep Onset measured by a polysomnograph | during the sleep time on the night(from 22:00-22:30 to the next morning wake-up)
Total sleep time measured by a polysomnograph | during the sleep time on the night(from 22:00-22:30 to the next morning wake-up)
Sleep efficiency measured by a polysomnograph | during the sleep time on the night(from 22:00-22:30 to the next morning wake-up)

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No